CLINICAL TRIAL: NCT00864864
Title: Pilot Study of Sunitinib Tumor Levels in Patients Not on Enzyme-Inducing Anti-Epileptic Drugs Undergoing Debulking Surgery for Recurrent Glioblastoma
Brief Title: Sunitinib Tumor Levels in Patients Not on Enzyme-Inducing Anti-Epileptic Drugs Undergoing Debulking Surgery for Recurrent Glioblastoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other); Dana-Farber Cancer Institute (Other); Pfizer (Industry)
Responsible Party: Principal Investigator, Scott Randall Plotkin, MD, PhD, Associate Professor of Neurology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-307
Record Dates: First submitted 2009-03-17; First posted 2009-03-19 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Glioblastoma; Brain Tumor
Keywords: sunitinib
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sunitinib (Experimental)
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — Taken orally on days 1-7 prior to surgery and then starting again on Day 22 for 4 weeks followed by a 2 week rest period

SUMMARY:
The purpose of this research study is to determine if sunitinib can get past the blood-brain barrier and into the brain tumor. Sunitinib has shown promising results in treating other cancers and works by blocking blood flow to tumors, which may prevent them from growing further. At the present time, there is no chemotherapy that can cure glioblastoma. The reason why chemotherapy is not fully effective is that many drugs cannot penetrate into brain tumors. This is due to the presence of the blood-brain barrier (BBB) which normally protects the brain from substances in the blood.

DETAILED DESCRIPTION:
* Participants will take the study drug, sunitinib, for 7 days prior to their surgery. The surgery is part of the routine care for glioblastoma and will be performed on Day 8. The study drug is supplied in capsule form and is to be taken at home.
* On Day 7 participants will come to the clinic and have the following tests and procedures performed: Neurological and physical examination; vital signs; and blood samples. On day 9 (the day after the surgery) an MRI scan will be performed.
* Fourteen days after the participants surgery (Day 22), they will restart sunitinib treatment. They will take the study drug once a day for 4 weeks followed by a 2 week rest period (no study drug treatment). This 6 week period is called a cycle of study treatment. Participants can continue to receive cycles of study treatment as long as their disease does not progress and they do not experience any serious side-effects.
* Before each new cycle of study treatment (once every 6 weeks) the participant will come into the clinic for the following tests: Neurological and physical examination; vital signs; blood sample; urine sample; MRI scan of the brain (done every even cycle).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed glioblastoma
* 18 years of age or older
* Karnofsky Performance Status 60 or greater
* Patient must be on no anti-epileptic drugs (AED) or AED that are non-enzyme inducing (NEIAED)
* There is no limit to the number of prior chemotherapy regimens
* No concurrent malignancy except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast. Patients with prior malignancies must be disease-free for 5 years or more
* Mini-mental status examination score of 15 or less
* Resolution of all acute toxic effect of prior chemotherapy, radiotherapy, or surgical procedures to grade 1 or less
* Adequate organ function as outlined in the protocol

Exclusion Criteria:

* Major surgery within 4 weeks of starting the study treatment
* Radiation therapy within 3 months of starting the study treatment
* Chemotherapy within 4 weeks (within 6 weeks for nitrosoureas) prior to entering the study
* Concurrent treatment on another clinical trial. Supportive care trials or non-treatment trials are allowed
* Any of the following within the 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure. stroke or transient ischemic attack, or pulmonary embolism
* Ongoing cardiac dysrhythmias of NCI CTCAE grade 2 or greater
* Prolonged QTc interval on baseline EKG
* Hypertension that cannot be controlled by medications
* Patients must not have a known coagulopathy that increases risk of bleeding or a history of clinically significant hemorrhages in the past
* Patients must be on therapeutic doses of anti-coagulants or anti-platelet agents while taking sunitinib
* Grade 3 systemic hemorrhage within 4 weeks fo starting the study treatment
* Patients whose MRI scan shows clinically significant intratumoral or peritumoral hemorrhage
* Pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness or active infection
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study
* Concomitant use of ketoconazole and other agents known to induce CYP3A4
* Pregnancy or breastfeeding
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to sunitinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-05; Primary Completion 2011-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
To assess the ability of sunitinib to achieve a target tumor: plasma ration greater than or equal to 0.2 in patients with recurrent GM. | 3 years

SECONDARY OUTCOMES:
To determine if there is an association between growth factor receptor inhibition and tumor phenotype, tumor: plasma ratio of sunitinib and overall survival. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Scott Plotkin, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts